CLINICAL TRIAL: NCT02158104
Title: Soreness After Deep Dry Needling of One Latent Myofascial Trigger Point
Status: Completed | Type: Observational
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Other Study IDs: CEU-004
Record Dates: First submitted 2014-06-05; First posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-01

CONDITIONS: Pain After Dry Needling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Latent trigger point in the upper trapezius muscle
  Interventions: Procedure: Deep dry needling

INTERVENTIONS:
Procedure: Deep dry needling

SUMMARY:
Pain after dry needling or injection in the muscle is a frequent secondary effect in the treatment of myofascial pain syndrome. In this trial pain and sensitivity will be assessed during a 72 hours follow up period. Factors that may contribute to higher levels of pain or sensitivity will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

The latent MTrP diagnosis was based upon the following criteria:10

1. presence of a palpable taut band in the muscle
2. presence of a hypersensitive tender spot in the taut band
3. palpable or visible local twitch response with snapping palpation of the tout band
4. referred pain elicitation in response to compression.

Exclusion Criteria:

1. presence of coagulation disorders
2. neck or facial pain
3. previous application of a dry needling technique
4. MTrP therapy in head or neck within the previous 3 months
5. fibromyalgia
6. an insurmountable fear of needles as a reason of refusing the treatment
7. history of surgery in the head or neck area.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjetct. Community sample from university.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Pain | 72 hours
  Visual analogue scale

SECONDARY OUTCOMES:
Sensitivity | 72 hours
  Pressure pain threshold